CLINICAL TRIAL: NCT04005040
Title: Evaluation of Mobile X-ray Within the Triple Aim Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Mobile X-ray
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2019-06

CONDITIONS: X-rays; Effects; Health Impairment; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Portable X-Ray

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: It is impossible to mask since patients are examined at the hospital or in their own home using mobile X-ray
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile X-ray (Active Comparator): Intervention: X-ray examination in the patients own home
  Interventions: Procedure: Mobile X-ray
- X-ray at the Hospital (Placebo Comparator): Control: X-ray at the hospital
  Interventions: Procedure: Mobile X-ray

INTERVENTIONS:
Procedure: Mobile X-ray — Evaluating the effect of mobile x-ray compared to x-ray at the Hospital

SUMMARY:
Background:

In foreign countries, mobile x-ray already is being used where transfer to the radiology department at the hospital may be an obstacle. Using mobile x-ray, the x-ray examination is performed in the patients own home with transportable equipment that reminds of the transportable x-ray equipment that is being used in the intensive care units. At The Department of Radiology (DOR), Aarhus University Hospital there is an ongoing project mobile x-ray for patients living in nursing homes in Aarhus. The project will be evaluated inspired by the Triple Aim Approach in three sub studies.

Overall aim:

The overall aim is to conclude if mobile x-ray improves healthcare for fragile patients.

Hypotheses:

* Patients examined with mobile x-ray have fewer number of hospital admissions compared with patients examined with x-ray at DOR.
* Patients examined with mobile x-ray are more satisfied with their examination compared with patients examined with x-ray at DOR.

Sub study 1 - Population health

Aim:

The primary aim is to study if mobile x-ray improves the health of the defined population measured in hospital admission. Also to study challenges conducting a RCT.

The outcome measures:

The primary outcome is hospital admissions.

Sub study 2 - Experience of care

Aim:

The aim is to study the satisfaction with mobile x-ray compared the satisfaction to x-ray at DOR.

Methods:

Observations, interview and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to a mobile X-ray examination in Aarhus Municipality

Exclusion Criteria:

* all other patients referred to an x-ray examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Hospital admissions | one year
  How many patients are hospitalized

SECONDARY OUTCOMES:
patient satisfaction | one year
  Measuring satisfaction using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Helene Nørrelund, Decan, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
The plan is not to share data with other reseachers

REFERENCES:
- [Result] Vigeland E, Bohm RE, Rostad A, Lysdahl KB. Mobile X-ray service for nursing homes. Tidsskr Nor Laegeforen. 2017 Feb 7;137(3):198-202. doi: 10.4045/tidsskr.16.0035. eCollection 2017 Feb. English, Norwegian. PMID 28181756